CLINICAL TRIAL: NCT02876406
Title: Using the ΔvapCO2 / Cav02 Ratio as a Prognostic Marker and Predictor of Complications After Cardiac Surgery
Brief Title: ΔvapCO2 / Cav02 Ratio as a Prognostic Marker and Predictor of Complications After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Tomás Francisco Fariña González, Resident Physician, Hospital San Carlos, Madrid
Other Study IDs: C.P. - C.I. 16/359-E
Record Dates: First submitted 2016-08-09; First posted 2016-08-23 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Surgery; Disorder of Blood Gas; Postoperative Complications; Shock
MeSH Terms: conditions — Postoperative Complications; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the usefulness of the ΔvapCO2 / Cav02 ratio to predict complications after elective cardiac surgery, comparing it with others markers such as lactate, arteriovenous CO2 difference (ΔvapCO2) and would try to developed a new predictive score for postoperative complications.

DETAILED DESCRIPTION:
Cardiac surgery is widely used to solve valvular or coronary problems and often requires the use of cardiopulmonary bypass or extracorporeal circulation (EC).

The EC itself produces a series of changes in the macro- and microcirculation hemodynamic and physiological consequences in the hours following surgery that can be difficult to analyze.

During postoperatively management, different monitoring methods are used to optimize different hemodynamic and analytical variables.

Sometimes, monitored variables are corrected but the patient still develops complications such as kidney failure, prolonged mechanical ventilation or even death. In fact, it is not well known either if it is sufficient to correct the variables called "macrodynamics " such as mean arterial pressure (MAP) , stroke volume (SV), pulmonary artery occlusion pressure (PCWP) and cardiac index (CI) or if it is necessary to correct other "micro-dynamics" variables like lactate, to achieve a certain central venous oxygen saturation (ScvO2) or arteriovenous CO2 difference(ΔvapCO2).

In tissue hypoxia, damping of excess protons by bicarbonate increase CO2 production; therefore the relationship between CO2 production and oxygen consumption (VCO2/VO2 ratio or respiratory quotient) increases. This ratio can be simplified relating ΔvapCO2 and O2 content arteriovenous difference (ΔvapCO2 / Cav02 ratio). In shock, anaerobic metabolism is one of the primary energy source. In this situation, ΔvapCO2 / Cav02 is > 1.

The evolution of the ΔvapCO2 / Cav02 ratio and its association with prognosis have nnot been studied yet after cardiac surgery.

The study's objectives are:

* to describe ΔvapCO2 / Cav02 ratios kinetics compared to lactate and other biochemical markers (troponin I, BE) in the first 12 hours after cardiac surgery.
* define if ΔvapCO2 / Cav02 ratio> 1 after 6 hours of adequate postsurgical resuscitation correlates with worse prognosis in patients after cardiac surgery.
* develop a new prognostic score for postoperative complication that includes ΔvapCO2 / Cav02 ratio.

Blood gases and drawn from a central venous and arterial lines. pCO2, O2 content, lactate are analyzed at 0, 2, 6 and 12 hs. Macrodynamic variables are also collected, as well as, the need of extracorporeal support techniques.

Patients would be followed for the next 28 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* given informed consent
* elective cardiac surgery
* tip of a central venous catheter correctly positioned (superior vena cava or right atria)
* arterial catheter correctly positioned

Exclusion criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery in an university hospital that would be followed during the postoperative time in the Cardiovascular Intensive Care Unit.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | within the first 28 days after surgery
all cause intra-ICU mortality | within the first 28 days after surgery
Ventilator days | within the first 28 days after surgery
  Time that is required to extubate the patient
ICU stay length | within the first 28 days after surgery
Hospital stay length | within the first 28 days after surgery
Acute kidney failure | within the first 28 days after surgery
  According RIFLE classification

SECONDARY OUTCOMES:
Vasoactive requirements after 12 hs | First 12 hs postoperative
  Noradrenaline or dobutamine requirement after 12 hs (yes/no)
Volume infused over 12 hs (ml) | First 12 hs postoperative
Intraaortic counterpulsation balloon | First 12 hs postoperative
  Need of Intraaortic baloon counterpulsation (yes/no)
Ventricular mechanical assistance | First 12 hs postoperative
  Need of ventricular mechanical assistance (yes/no)
Renal replacement therapies | within the first 28 days after surgery
  Need of renal replacement therapies (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du W, Long Y, Wang XT, Liu DW. The Use of the Ratio between the Veno-arterial Carbon Dioxide Difference and the Arterial-venous Oxygen Difference to Guide Resuscitation in Cardiac Surgery Patients with Hyperlactatemia and Normal Central Venous Oxygen Saturation. Chin Med J (Engl). 2015 May 20;128(10):1306-13. doi: 10.4103/0366-6999.156770. PMID 25963349
- [Background] Hu BY, Laine GA, Wang S, Solis RT. Combined central venous oxygen saturation and lactate as markers of occult hypoperfusion and outcome following cardiac surgery. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):52-7. doi: 10.1053/j.jvca.2011.07.021. Epub 2011 Sep 15. PMID 21924630
- [Background] Habicher M, von Heymann C, Spies CD, Wernecke KD, Sander M. Central Venous-Arterial pCO2 Difference Identifies Microcirculatory Hypoperfusion in Cardiac Surgical Patients With Normal Central Venous Oxygen Saturation: A Retrospective Analysis. J Cardiothorac Vasc Anesth. 2015;29(3):646-55. doi: 10.1053/j.jvca.2014.09.006. Epub 2015 Jan 6. PMID 25575410
- [Background] Robin E, Futier E, Pires O, Fleyfel M, Tavernier B, Lebuffe G, Vallet B. Central venous-to-arterial carbon dioxide difference as a prognostic tool in high-risk surgical patients. Crit Care. 2015 May 13;19(1):227. doi: 10.1186/s13054-015-0917-6. PMID 25967737
- [Background] Mekontso-Dessap A, Castelain V, Anguel N, Bahloul M, Schauvliege F, Richard C, Teboul JL. Combination of venoarterial PCO2 difference with arteriovenous O2 content difference to detect anaerobic metabolism in patients. Intensive Care Med. 2002 Mar;28(3):272-7. doi: 10.1007/s00134-002-1215-8. Epub 2002 Feb 8. PMID 11904655
- [Background] Ospina-Tascon GA, Umana M, Bermudez W, Bautista-Rincon DF, Hernandez G, Bruhn A, Granados M, Salazar B, Arango-Davila C, De Backer D. Combination of arterial lactate levels and venous-arterial CO2 to arterial-venous O 2 content difference ratio as markers of resuscitation in patients with septic shock. Intensive Care Med. 2015 May;41(5):796-805. doi: 10.1007/s00134-015-3720-6. Epub 2015 Mar 20. PMID 25792204
- [Background] Balzer F, Sander M, Simon M, Spies C, Habicher M, Treskatsch S, Mezger V, Schirmer U, Heringlake M, Wernecke KD, Grubitzsch H, von Heymann C. High central venous saturation after cardiac surgery is associated with increased organ failure and long-term mortality: an observational cross-sectional study. Crit Care. 2015 Apr 16;19(1):168. doi: 10.1186/s13054-015-0889-6. PMID 25888321